CLINICAL TRIAL: NCT05727007
Title: Evaluation of Computed Tomography and Magnetic Diffusion Resonance Imaging in the Preoperative Staging of Colon Cancer
Brief Title: CT and MRI in Preoperative Colon Cancer Staging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Effrosyni Bompou, Effrosyni Bompou Principal Investigator, Larissa University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTMR
Record Dates: First submitted 2023-01-25; First posted 2023-02-14 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Colonic Neoplasms
Keywords: colon; cancer; computed tomography; magnetic resonance; diffusion; preoperative; staging
MeSH Terms: conditions — Colonic Neoplasms; Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: The study will employ a prospective design
Masking Description: There will be no blindness at the level of the patient, the treating physicians (surgeon, oncologist, radiologist) and the researcher who will record the data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI in colon cancer (Experimental): All prospectively included patients with colon cancer will be preoperatively submitted to MRI for staging. The evaluation of the diagnostic accuracy will be based on the cross-examination with the CT scan and the pathology results
  Interventions: Diagnostic Test: MRI in colon cancer; Diagnostic Test: CT in colon cancer

INTERVENTIONS:
Diagnostic Test: MRI in colon cancer — The MRI protocol will include the following imaging series: T1 and T2 in axial and coronal plane before the administration of intravenous contrast, diffuse weight imaging in axial plane and T1 after the administration of intravenous contrast
Diagnostic Test: CT in colon cancer — The CT scan protocol will include the following: per os and intravenous administration of contrast, axial slices of 0.3mm thickness and reconstruction per 1mm, multi-planar reformation and three-dimensional volume rendering

SUMMARY:
The objective of this study is the evaluation of different imaging methods for the optimal preoperative staging of colon cancer patients. Imaging findings will be compared with the histopathologic results of the specimen following surgical resection.

DETAILED DESCRIPTION:
Over the last years a significant improvement in the treatment of patients with colon cancer has been reported. This has been attributed to the improvement of the staging techniques, as well as the optimization of the surgical management. However, the current five-year survival rates of colon cancer patients in European countries ranges from 32% to 64%. This variation could be due to treatment discrepancies and the lack of adherence to the international guidelines.

Surgical treatment of colon cancer includes the radical resection of the tumour (colectomy). Following resection, the specimen is histopathologically examined, the disease is staged and further treatment is determined. Neoadjuvant treatment (radiotherapy or/and chemotherapy) for colon cancer has not been yet approved, unlike rectal cancer, where neoadjuvant treatment is recommended for specific disease stages.

Preoperative staging of colon cancer aims to identify those patients with remote metastatic disease, who will, more likely, not benefit from upward surgery. Recent developments in colon cancer management, demanding more precise local disease staging, to identify those patients who will likely benefit from neoadjuvant chemotherapy, are still at a clinical trial stage.

Preoperative treatment depends on the disease stage, which is defined by the tumour's invasion in the colonic wall, the dissemination in nearby organs or lymph nodes, and the presence of distal metastases. The stage is first evaluated radiologically and then confirmed via histopathological examination of the specimen. Imaging is an already approved tool for the staging of colonic cancer, while in some studies the combination of different imaging methods has been reported to improve the initial evaluation.

Over the last years, evaluation of the circumferential resection margin (CRM) is also recommended in the preoperative staging of patients with colon cancer. This assessment is particularly important for tumours located at the cecum, right, or left colon, since these areas lack of mobile mesocolon and therefore it is possible to infiltrate the retroperitoneal resection margin.

Nevertheless, the retroperitoneal invasion of these tumours has not been evaluated adequately as a preoperative marker for both local recurrence and for the selection of patients who may benefit from neoadjuvant treatment. In various studies the percentage of retroperitoneal resection margin's infiltration was between 7-10% for cecum and right colon adenocarcinomas, while its presence was identified as a risk factor for local recurrence. The retroperitoneal surface infiltration was preoperatively evaluated with the combination of imaging methods and the findings were postoperatively compared with the histopathological features of the specimen.

A more precise, imaging based, preoperative staging, could lead to a more targeted neoadjuvant treatment for patients with advanced disease, with the introduction of chemo- and/or radiotherapy. This approach could result to the downstaging of the tumour, with better short and long term oncological results.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colonic adenocarcinoma
* Patient 18 to 90 years old
* Abscence of comorbidities that may affect treatment
* Signed informed consent of the patient

Exclusion Criteria:

* Inability to receive or contraindication for intravenous contrast
* Renal impairment
* Previous allergies to intravenous contrasts
* Incompatible implants with magnetic resonance imaging
* Claustrophobia
* Active sepsis or systemic infection
* Untreated physical and mental disability
* Lack of compliance with the protocol process
* Non-granting of signed informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy in T stage | 1 month postoperatively
  Evaluation of diagnostic accuracy in the T stage assessment. Diagnostic accuracy will be evaluated in terms of specificity (true negative rate)

SECONDARY OUTCOMES:
Diagnostic accuracy in N stage | 1 month postoperatively
  Evaluation of diagnostic accuracy in the presence of local or distant metastatic lymph nodes. Diagnostic accuracy will be evaluated in terms of specificity (true negative rate)
Diagnostic accuracy in the retroperitoneal resection margin | 1 month postoperatively
  Evaluation of diagnostic accuracy in the retroperitoneal resection margin. Diagnostic accuracy will be evaluated in terms of specificity (true negative rate)
Diagnostic accuracy in peritoneal or nearby organ infiltration | 1 month postoperatively
  Evaluation of diagnostic accuracy in the peritoneal or nearby organ infiltration. Diagnostic accuracy will be evaluated in terms of specificity (true negative rate)

CONTACTS AND LOCATIONS:
Overall Officials: George Tzovaras, Prof, Study Chair — University Hospital of Larissa; Effrosyni Bompou, MSc, Principal Investigator — University Hospital of Larissa
Locations (1):
- Department of Surgery, University Hospital of Larissa, Larissa, Greece

IPD SHARING:
Plan to Share IPD: No
No plan to share individual patient data

REFERENCES:
- [Background] Xynos E, Gouvas N, Triantopoulou C, Tekkis P, Vini L, Tzardi M, Boukovinas I, Androulakis N, Athanasiadis A, Christodoulou C, Chrysou E, Dervenis C, Emmanouilidis C, Georgiou P, Katopodi O, Kountourakis P, Makatsoris T, Papakostas P, Papamichael D, Pentheroudakis G, Pilpilidis I, Sgouros J, Vassiliou V, Xynogalos S, Ziras N, Karachaliou N, Zoras O, Agalianos C, Souglakos J; [the Executive Team on behalf of the Hellenic Society of Medical Oncology (HeSMO)]. Clinical practice guidelines for the surgical management of colon cancer: a consensus statement of the Hellenic and Cypriot Colorectal Cancer Study Group by the HeSMO. Ann Gastroenterol. 2016 Jan-Mar;29(1):3-17. PMID 26752945
- [Background] Nelson H, Petrelli N, Carlin A, Couture J, Fleshman J, Guillem J, Miedema B, Ota D, Sargent D; National Cancer Institute Expert Panel. Guidelines 2000 for colon and rectal cancer surgery. J Natl Cancer Inst. 2001 Apr 18;93(8):583-96. doi: 10.1093/jnci/93.8.583. PMID 11309435
- [Background] Jhaveri KS, Hosseini-Nik H. MRI of Rectal Cancer: An Overview and Update on Recent Advances. AJR Am J Roentgenol. 2015 Jul;205(1):W42-55. doi: 10.2214/AJR.14.14201. PMID 26102418
- [Background] Foxtrot Collaborative Group. Feasibility of preoperative chemotherapy for locally advanced, operable colon cancer: the pilot phase of a randomised controlled trial. Lancet Oncol. 2012 Nov;13(11):1152-60. doi: 10.1016/S1470-2045(12)70348-0. Epub 2012 Sep 25. PMID 23017669
- [Background] Nerad E, Lambregts DM, Kersten EL, Maas M, Bakers FC, van den Bosch HC, Grabsch HI, Beets-Tan RG, Lahaye MJ. MRI for Local Staging of Colon Cancer: Can MRI Become the Optimal Staging Modality for Patients With Colon Cancer? Dis Colon Rectum. 2017 Apr;60(4):385-392. doi: 10.1097/DCR.0000000000000794. PMID 28267005
- [Background] Jacobs MA, Macura KJ, Zaheer A, Antonarakis ES, Stearns V, Wolff AC, Feiweier T, Kamel IR, Wahl RL, Pan L. Multiparametric Whole-body MRI with Diffusion-weighted Imaging and ADC Mapping for the Identification of Visceral and Osseous Metastases From Solid Tumors. Acad Radiol. 2018 Nov;25(11):1405-1414. doi: 10.1016/j.acra.2018.02.010. Epub 2018 Apr 4. PMID 29627288
- [Background] Kijima S, Sasaki T, Nagata K, Utano K, Lefor AT, Sugimoto H. Preoperative evaluation of colorectal cancer using CT colonography, MRI, and PET/CT. World J Gastroenterol. 2014 Dec 7;20(45):16964-75. doi: 10.3748/wjg.v20.i45.16964. PMID 25493009
- [Background] Antoch G, Vogt FM, Freudenberg LS, Nazaradeh F, Goehde SC, Barkhausen J, Dahmen G, Bockisch A, Debatin JF, Ruehm SG. Whole-body dual-modality PET/CT and whole-body MRI for tumor staging in oncology. JAMA. 2003 Dec 24;290(24):3199-206. doi: 10.1001/jama.290.24.3199. PMID 14693872
- [Background] Hunter C, Blake H, Jeyadevan N, Abulafi M, Swift I, Toomey P, Brown G. Local staging and assessment of colon cancer with 1.5-T magnetic resonance imaging. Br J Radiol. 2016 Aug;89(1064):20160257. doi: 10.1259/bjr.20160257. Epub 2016 May 26. PMID 27226219
- [Background] Ellebaek SB, Fristrup CW, Mortensen MB. Intraoperative Ultrasound as a Screening Modality for the Detection of Liver Metastases during Resection of Primary Colorectal Cancer - A Systematic Review. Ultrasound Int Open. 2017 Apr;3(2):E60-E68. doi: 10.1055/s-0043-100503. Epub 2017 Jun 7. PMID 28597000
- [Background] Elibol FD, Obuz F, Sokmen S, Terzi C, Canda AE, Sagol O, Sarioglu S. The role of multidetector CT in local staging and evaluation of retroperitoneal surgical margin involvement in colon cancer. Diagn Interv Radiol. 2016 Jan-Feb;22(1):5-12. doi: 10.5152/dir.2015.15089. PMID 26611110
- [Background] Bateman AC, Carr NJ, Warren BF. The retroperitoneal surface in distal caecal and proximal ascending colon carcinoma: the Cinderella surgical margin? J Clin Pathol. 2005 Apr;58(4):426-8. doi: 10.1136/jcp.2004.019802. PMID 15790712
- [Background] Hajian-Tilaki K. Sample size estimation in diagnostic test studies of biomedical informatics. J Biomed Inform. 2014 Apr;48:193-204. doi: 10.1016/j.jbi.2014.02.013. Epub 2014 Feb 26. PMID 24582925
- [Background] Heald RJ, Husband EM, Ryall RD. The mesorectum in rectal cancer surgery--the clue to pelvic recurrence? Br J Surg. 1982 Oct;69(10):613-6. doi: 10.1002/bjs.1800691019. PMID 6751457
- [Background] West NP, Hohenberger W, Weber K, Perrakis A, Finan PJ, Quirke P. Complete mesocolic excision with central vascular ligation produces an oncologically superior specimen compared with standard surgery for carcinoma of the colon. J Clin Oncol. 2010 Jan 10;28(2):272-8. doi: 10.1200/JCO.2009.24.1448. Epub 2009 Nov 30. PMID 19949013

DOCUMENTS (2):
  • Study Protocol (2023-01-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT05727007/Prot_000.pdf
  • Informed Consent Form (2023-01-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT05727007/ICF_001.pdf